CLINICAL TRIAL: NCT04913558
Title: Effect of Aerobic Exercise on Stress and Fatigue of Lactating Employed Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Elsayed Basyouny Zaher, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sarazaher_Msc
Record Dates: First submitted 2021-05-29; First posted 2021-06-04 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Stress; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Treatment Arm (Active Comparator): This group will consist of thirty employed lactating women suffering from stress and fatigue. This group will receive the same lifestyle modification advice that will be given to the aerobic exercise group during the six weeks of the program period.
  Interventions: Other: Traditional Treatment
- Aerobic exercise group (Experimental): This group will consist of thirty employed lactating women suffering from stress and fatigue. These women will perform aerobic exercise for 30 minutes for each session, 5 times per week, for 6 weeks in the form of treadmill training (60- 70% of HR max) and do some modifications of their routine by following lifestyle modification advice given to them during the 6 weeks of the program period.
  Interventions: Other: Aerobic exercise; Other: Traditional Treatment

INTERVENTIONS:
Other: Aerobic exercise — The exercise will be performed by using the treadmill as the following:
  - The first stage (warming up): It consists of 5 minutes warming up with the treadmill speed set at 1.0 mile per hour.
  - The second stage (active stage): It consists of 20 minutes with the treadmill speed set at 3.0 miles per hour.
  - Third stage (cooling down): It consists of 5 minutes of cooling down with the treadmill speed set at 1.0 miles per hour.
  Arms: Aerobic exercise group
Other: Traditional Treatment — 1. General advice for reducing fatigue and stress
  2. Fluid and diet advice
  3. Carrying the Baby
  4. While Breastfeeding in a sitting position
  5. Selecting Clothing

SUMMARY:
The study aims to determine the effect of aerobic exercise on stress and fatigue of employed lactating women.

DETAILED DESCRIPTION:
The study aims to determine the effect of aerobic exercise on stress and fatigue of employed lactating women. This study will be carried out on Sixty lactating mothers working in the medical field who have returned to work after maternity leave and suffering from stress and fatigue.

The subjects will be divided randomly into two groups equal in number, the Aerobic exercise group ( group A) and the Control group ( group B).

Group A will consist of thirty employed lactating women suffering from stress and fatigue. These women will perform aerobic exercise for 30 minutes for each session, 5 times per week, for 6 weeks in the form of treadmill training (60- 70% of HR max) and do some modifications of their routine by following lifestyle modification advice given to them during the 6 weeks of the program period.

Control group (group B):

This group will consist of thirty employed lactating women suffering from stress and fatigue. This group will receive the same lifestyle modification advice that will be given to group (A) during the six weeks of the program period.

ELIGIBILITY:
Inclusion Criteria:

* All participants are lactating mothers.
* Working in the medical field 4 to 6 hours per day, 4 to 5 days per week.
* Returned to work after 4 months of maternity leave.
* Suffering stress and fatigue considering the perceived stress questionnaire and the fatigue assessment scale.
* Their babies' ages will be ranged from 6 to 8 months old.
* Having at least one year of work experience before giving birth.
* Their age will be ranged from 25 to 35 years.
* They haven't exercised more than twice per week during the previous 3 months.

Exclusion Criteria:

* Any neurological, cardiovascular disorders, or metabolic disease
* Physical impairments that prevent following the program.
* Women who are planning to stop breastfeeding in the next 4 months.
* Women with regular medications.
* Mothers of formula feeding babies.
* women who are smoking will be excluded from this study.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — lactating mothers working in the medical field who have returned to work after maternity leave and suffering from stress and fatigue.
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Stress assessment | Baseline and 6 weeks post-intervention
  Change from baseline of stress at 6 weeks. Assessment of stress through using perceived stress scale 10 will be performed before and after intervention
Fatigue assessment | Baseline and 6 weeks post-intervention
  Change from baseline of stress at 6 weeks. Assessment of fatigue through using fatigue assessment scale will be performed before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sara Zahrer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No